CLINICAL TRIAL: NCT04935671
Title: Co-administration of Saffron and Chamomile: to Determine the Efficacy as an Adjuvant Therapy for Mild to Moderate Depression in Human Subjects
Brief Title: Effects of Saffron and Chamomile in Mild to Moderate Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr Saara (Ahmad) Muddasir Khan (Other)
Collaborators: University of Karachi (Other)
Responsible Party: Sponsor-Investigator, Dr Saara (Ahmad) Muddasir Khan, Assistant Professor, Aga Khan University
Organization: Aga Khan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0924
Record Dates: First submitted 2021-05-31; First posted 2021-06-23 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Depression
Keywords: Depression; Diabetes; PHQ9; saffron; chamomile
MeSH Terms: conditions — Depression; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study design will be prospective, randomized, open-labeled, blinded end-point trial for a period of 4-weeks.
Who Masked: Outcomes Assessor
Masking Description: blocked randomization technique has done via software
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allopathic + Herbal (Active Comparator): 20mg of chamomile and 1 mg saffron in form of teabag for preparation of herbal decoction in dose of two teabags per day for a month as an "ADJUVANT THERAPY" with standard allopathic treatment for depression.
  Interventions: Dietary Supplement: chamomile tea n saffron
- Allopathic only (No Intervention): Only allopathic medication for depression.

INTERVENTIONS:
Dietary Supplement: chamomile tea n saffron — 20 mg of chamomile and 1 mg saffron in a teabag given twice daily for a month in combination with allopathic treatment for depression.
  Arms: Allopathic + Herbal

SUMMARY:
Diabetes characterized by decreased production, or resistance to the action of insulin or both. The reduced production or action alters many important body functions namely glucose absorption and utilization in the body. The disturbed glucose metabolism profoundly effects transportation of large neutral amino acids especially tryptophan in brain leading decreased synthesis of serotonin and hence ensuing depression, memory loss and various other psycho-neurological problems.

Different antipsychotic treatments like serotonin reuptake inhibitors, monoamine inhibitors and tricyclic antidepressants are available in the market to treat depression but are not devoid of adverse effects. Therefore, there is a tendency in underdeveloped countries to use alternative remedies to combat the psycho-neurological issues. Nature has bestowed the bounty of indigenous herbs like Saffron (Crocus sativusL) and chamomile (Matricaria chamomileL), that possess neuro-protective effects and are regularly consumed in day to day delicacies with no documented adverse-effects nor adverse events Though these herbs have been studied widely for their multiple therapeutic benefits, however, till date both of these herbs in combination have not been studied as an adjuvant therapy for mild to moderate depression. Therefore the present study is designed to determine the combined beneficial effects of these herbs as an adjuvant therapy for treatment of depression.

DETAILED DESCRIPTION:
Depression is a psychological state constellation of sad mood, agitation, lack of interest and feelings of worthlessness. Depression may be developed or aggravated by multiple factors like death of a loved one, unhealthy living environmental condition, seasonal variations and during postpartum state. It has been studied previously that the brain neurotransmitters, monoamines namely serotonin, dopamine and/or norepinephrine are altered in depression. The most notable monoamine that plays a vital role is serotonin also known as 5 hydroxy tryptamine (5- HT). The precursor of serotonin in brain is identified as tryptophan and its transport in brain declines leading to reduced synthesis of serotonin and hence ensuing depressive states. It is also noted that serotonin production is decreased profoundly in diabetic subjects. Insulin plays a vital role in mobilization of tryptophan into brain by facilitating transport of other large neutral amino acids in somatic compartments. Hence, insulin resistance or its deficiency leads to compromised access of tryptophan in the brain ultimately resulting in reduced production of serotonin causing depression.

Likewise the composition of diet consumed does have a major role in the mood alteration. Upon consumption of protein rich food, the concentrations of large neutral amino acids levels are increased in the blood. The competition between the large neutral amino acids and the tryptophan at the brain receptor level to cross the blood brain barrier increases leading to relatively lesser transport of tryptophan in the brain. On the other hand, food rich in carbohydrates in normo-glycemics causes increase sugar levels in the blood resulting in increased insulin secretion. The optimal level of insulin enhances the entry of large neutral amino acids in the body tissues leaving increased tryptophan to enter brain.

The prevalence of depression in the population Karachi, Pakistan is known to be 25- 30%. Different antipsychotic treatments like serotonin reuptake inhibitors, monoamine inhibitors and tricyclic antidepressants are commonly available in the market to treat anxiety and depression. Their principle action is mediated through alteration of the brain neurotransmitters levels, however, their short and/or long term administration may precipitate wide range of adverse effects including tolerance and habituation, insomnia, suicidal tendency and aggravation of depressive episodes. Therefore, there is a popular trend in developing countries to use alternative remedies for the treatment of psycho-neurological issues like depression and nature has bestowed the bounty of indigenous herbs that possess neuro-protective effects and may be used for medicinal purpose in population. Crocus sativusL. commonly known as Saffron and Matricaria chamomileL. referred as chamomile, have been used since ages for the diverse medicinal benefits such as fever, inflammation, muscle spasms, menstrual disorders, infertility, gastric ulcers, insomnia, depression, anxiety and dementia. These herbs are regularly consumed in day to day delicacies and have largely been found safe at tolerated dose ranges.

Saffron The main components of saffron are crocin, picrocrocin and safranal. The median lethal doses (LD50) of saffron are 200 mg/ml and 20.7 g/kg in vitro and in animal studies, respectively. Saffron has been suggested to be effective in the treatment of a wide range of disorders including coronary artery diseases, hypertension, stomach disorders, dysmenorrhea and depression, anxiety, learning and memory impairments. Saffron is reported to be effective for depression at 30mg/kg/oral dose or in two divided doses of 15 mg/kg body weight, while its higher doses (200-800 mg/kg body weight) administered orally were found to be effective for the treatment of epilepsy and Alzheimer's disease. Similarly, diverse dose-range has been used for the treatment of asthma, cough, hemoptysis, Alzheimer's disease, heart burn, infertility, PCOS, anti-inflammatory, anti-sclerotic as well as neuro-protective agent. Administration of saffron and its constituents increases glutamate and dopamine levels in the brain. It has also demonstrated antidepressant effects in clinical studies and extensive anxiolytic effects in experimental animal models.

Likewise, chamomile has also demonstrated neuro-protective and anxiolytic effects in the both human and animal model.

Chamomile The main components of chamomile are bisabolo. The median lethal doses (LD50) of chamomile are 15ml/kg. However, 1-2 ml/ kg of bisabolol can be well tolerated by rats. Chamomile has been found well found well tolerated up to the dose of 1500 mg/kg/day with no severe adverse effects. Chamomile is reported to be effective in the dose range from 30 mg/kd/day to 100mg/kg/day in form of ethanolic extract or water decoction. Different dose ranges are used for the treatment of various ailments like 9-15g/kg/day for respiratory infections, 30mg/kg/day to 100mg/kg/day for the treatment of eczema, skin infections, and Chrons disease, abdominal spasm, diarrhea, infertility, in post-menopausal states, respiratory and renal infections and inflammations as well as mood swings and anxiety. Several lines of evidence suggest that most of the flavonoid constituents of chamomile may produce anxiolytic activity by affecting γ-amino butyric acid (GABA), noradrenalin (NA), dopamine (DA), and serotonin neurotransmission or by modulating hypothalamic-pituitary-adrenocortical axis function.

Though there are studies are available in literature supporting the clinical efficacy of saffron or chamomile in anxiety or depression, there is no single study highlighting the potential benefits of co-administration of saffron and chamomile tea for the treatment of mild to moderate depression with or without co-morbid diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to moderate depression
* tea bags for preparation of herbal decoction will be given as adjuvant therapy

Exclusion Criteria:

* cancer
* morbid depression

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Depression | 1 month
  100 participants with adjuvant therapy in Arm A (allopathic+herbal) and 100 participants of Arm B with allopathic treatment only will be assessed by PHQ 9 questionnaire before and after intervention through change in PHQ 9 score.

SECONDARY OUTCOMES:
Glucose | 1 month
  the concentration of glucose will be measured in all participants for normoglycemia (fasting glucose: 65-100mg/dl) before and after intervention.
lipid profile | 1 month
  the concentration of lipids (serum cholesterol 200mg/dl, triglycerides <150mg/dl, HDL-cholesterol >40mg/dl, LDL-cholesterol<100mg/dl, VLDL-cholesterol <100mg/dl) will be measured in all participants before and after intervention.
Tryptophan | 1 month
  the level of tryptophan (0.34-80 ng/mL) will be measured in all participants before and after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, PK, Pakistan